CLINICAL TRIAL: NCT02024373
Title: Multi-Center, Randomized, Placebo-Controlled, Double Blind Study of the Atorvastatin: Effect on Patients With Chronic Subdural Hematoma
Brief Title: Effect and Safety Study of Atorvastatin to Treat Chronic Subdural Hematoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oriental Neurosurgery Evidence-Based-Study Team (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSDH2013
Record Dates: First submitted 2013-08-07; First posted 2013-12-31 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Subdural Hematoma
Keywords: chronic subdural hematoma; Atorvastatin; oral administration therapy
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental): atorvastatin：20 mg (every evening orally) for 8 weeks
  Interventions: Drug: Atorvastatin
- placebo (Placebo Comparator): placebo:20 mg (every evening orally) for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Atorvastatin — 20 mg (every evening orally) for 8 weeks
  Arms: Atorvastatin
Drug: placebo — 20 mg (every evening orally) for 8 weeks
  Arms: placebo

SUMMARY:
To evaluate the clinic effects and security of oral administration of Atorvastatin on chronic subdural hematoma (CSDH).

DETAILED DESCRIPTION:
Study design:

Multi-center, randomized, double-blind, placebo parallel controlled

Subjects:

Patients with chronic subdural hematoma (CSDH)

Sample size:

200, including an Atorvastatin-treated group of 100 patients and a control group of 100 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and <90 years old, male or female;
2. CT scan reveals supratentorial, unilateral or bilateral chronic subdural hematoma (MRI scan is warranted if diagnosis is difficult);
3. Markwalder's Grading Scale and Glasgow Coma Scale (MGS-GCS)<Grade 3;
4. Attending physician makes a judgment that cerebral hernia would not occur and surgical operation might not be performed in a short time. Conservative treatment is adopted;
5. Patients have never undergo surgery on the hematoma
6. Patient fully understood the nature of the study, and voluntarily participates and signs informed consent.

Exclusion Criteria:

1. Allergic to the statin or its ingredients
2. Cerebral herniation might occur at any time;
3. Hematoma leads to herniation and warrants surgical operation.
4. Hematoma caused by tumors, blood and other known comorbidities;
5. Abnormal liver function
6. Uncontrolled hepatitis and other liver diseases, as well as suffering from other disease may interfere the study
7. Patients have been on oral Statin treatment for a long time.
8. Patients have been on oral Steroids treatment for a long time.
9. Participate in clinical trials in the past four weeks;
10. Pregnant or breastfeeding
11. Failure of completing the trial by poor compliance;
12. For any reason, the researchers believe that the case is not suitable for inclusion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-12; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Hematoma Reduced Amount. | Check on 8 weeks during treatment (at the end)
  The primary efficacy endpoint: hematoma reduced amount. Outcome Measures: all patients underwent head CT (plain scan) before treatment, and check on 8 weeks during treatment (at the end)

SECONDARY OUTCOMES:
The consciousness score (MGS-GCS) and outcome score (GOS, ADL-BI Scale) in subjects | 0，7days，4, 8weeks during treatment (at the end), in the follow-up in 12 and 24 weeks.
Changes of neurological symptoms and signs | 0，7days，4, 8weeks during treatment (at the end), in the follow-up in 12 and 24 weeks.
Changes of routine blood test and coagulation results | 0，7days，4, 8weeks during treatment (at the end), in the follow-up in 12 and 24 weeks.
Hematoma Reduced Amount | 4 weeks during treatment, in the follow-up in 12 and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ning jian zhang, MD, PhD, Principal Investigator — Tianjin Medical University General Hospital
Locations (31):
- China (31):
  - Beijing tiantan hospital, Beijing, Beijing Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Chinese PLA General Hospital, Beijing
  - Peking union medical college hospital, Beijing
  - Cangzhou centerl hospital, Cangzhou
  - Xiangya hospital central southe university, Changsha
  - Southwest hospital, Chongqing
  - West china hospital, Chongqing
  - The first affiliated hospital of Fujian medical university, Fuzhou
  - Nanfang hospital, Guangzhou
  - First Affiliated Hospital of Harbin Medical University, Haerbing
  - Hainan general hospital, Haikou
  - 117 Hospital of People's Liberation Army, Hangzhou
  - The second Affiliated hospital of zhejiang university school of medicine, Hangzhou
  - Anhui provincial hospital, Hefei
  - Inner mongolia people's hospital, Hohehot
  - Qilu hospital of shandong university, Jinan
  - Linyi People's Hospital, Linyi
  - Jiangsu province hospital, Nanjing
  - Ordos Central Hospital, Ordos
  - Changzheng Hospital, Shanghai
  - Huashan hospital, Shanghai
  - The second hospital of Hebei medical university, Shijiazhuang
  - The first hospital of Shanxi medical university, Taiyuan
  - Tongji hospital, Wuhan
  - Tangdu hospital, Xi'an
  - Xijing Hospital, Xi'an
  - Prince of Wales Hospital, Xianggang
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - General Hospital of Ningxia Medical University, Yinchuan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

REFERENCES:
- [Derived] Wang D, Tian Y, Wei H, Gao C, Fan Y, Yang G, Quan W, Huang J, Yue S, Zhang J, Jiang R. Risk Factor Analysis of the Conservative Treatment in Chronic Subdural Hematomas: A Substudy of the ATOCH Trial. Adv Ther. 2022 Apr;39(4):1630-1641. doi: 10.1007/s12325-022-02057-w. Epub 2022 Feb 8. PMID 35133631
- [Derived] Jiang R, Zhao S, Wang R, Feng H, Zhang J, Li X, Mao Y, Yuan X, Fei Z, Zhao Y, Yu X, Poon WS, Zhu X, Liu N, Kang D, Sun T, Jiao B, Liu X, Yu R, Zhang J, Gao G, Hao J, Su N, Yin G, Zhu X, Lu Y, Wei J, Hu J, Hu R, Li J, Wang D, Wei H, Tian Y, Lei P, Dong JF, Zhang J. Safety and Efficacy of Atorvastatin for Chronic Subdural Hematoma in Chinese Patients: A Randomized ClinicalTrial. JAMA Neurol. 2018 Nov 1;75(11):1338-1346. doi: 10.1001/jamaneurol.2018.2030. PMID 30073290
- [Derived] Jiang R, Wang D, Poon WS, Lu YC, Li XG, Zhao SG, Wang RZ, You C, Yuan XR, Zhang JM, Feng H, Fei Z, Yu XG, Zhao YL, Hu J, Kang DZ, Yu RT, Gao GD, Zhu XD, Sun T, Hao JH, Liu XZ, Su N, Yue SY, Zhang JN. Effect of ATorvastatin On Chronic subdural Hematoma (ATOCH): a study protocol for a randomized controlled trial. Trials. 2015 Nov 18;16:528. doi: 10.1186/s13063-015-1045-y. PMID 26581842